CLINICAL TRIAL: NCT02059395
Title: Mastery Learning Versus Time-based Education: Skill Acquisition and Retention of Basic Life Support in Laypeople
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Mastery of BLS
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2017-03

CONDITIONS: Basic Life Support; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Time based (Active Comparator): Participants follow the traditional Canadian Heart and Stroke Foundation Heartsaver Course
  Interventions: Other: Time based learning
- Mastery based (Experimental): Participants do follow the content of the Canadian Heart and Stroke Foundation Heartsaver Course content based on their own pace (timeframe)
  Interventions: Other: Mastery based learning

INTERVENTIONS:
Other: Mastery based learning — Participants are allowed to follow the course content at their own speed
  Arms: Mastery based
Other: Time based learning — Participants follow the traditional Canadian Heart and Stroke Foundation Heartsaver Course according to the official course layout
  Arms: Time based

SUMMARY:
Background:

In cardiac arrest survival rates dramatically increase when bystanders are present and initiate Basic Life Support (BLS). However, even though serious efforts have been made, skill retention after a traditional time-based BLS course for laypeople remains suboptimal. In contrast, a mastery learning-based educational approach was shown to be efficacious and might be promising even for laypersons. Therefore the investigators aim to evaluate the impact of a mastery learning-based BLS course on skills retention of BLS in laypeople.

Methods:

Forty laypeople without previous BLS experiences will be randomized into the traditional time-based BLS course group (Control - TB group) or mastery learning-based group (Intervention - ML group).

Both groups will receive BLS training consisting of 6 successive stations including diagnosis of cardiac arrest, chest compression, ventilation, one-rescuer BLS, two-rescuer BLS and AED use. In the ML group, subjects will deliberately practice and receive feedback at each station until a pre-set target level is reached. Subjects will be allowed to proceed to the next station only when they achieve the required target level of performance. In contrast, participants of the TB group will be taught the same 6 stations in two hours, according to standard American Heart Association BLS criteria. All subjects will have an assessment of knowledge and skills immediately after teaching (immediate post-test) and at four months (retention post-test).

Implications:

Previous research has shown that mastery learning-based education improves learners' procedural skill performance. The investigators study will determine the impact of a mastery learning-based BLS course on skill retention in laypeople.

ELIGIBILITY:
Inclusion Criteria:

* University students in Ottawa

Exclusion Criteria:

* Students of the Faculty of Medicine
* Previous Basic Life Support Training Certificate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2015-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Boet, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The University of Ottawa Skills and Simulation Centre, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Time Based | Mastery Based
Started | 22 | 27
Completed | 20 | 23
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Time Based | Mastery Based | Total
Number analyzed (Participants) | 22 | 27 | 49
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 19.5 [18.0 to 21.0] | 20.0 [18.75 to 21.0] | 19.7 [18.5 to 21.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 13 | 14 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Skill Retention Estimated From the Change of AHA Heartsaver Total Score From Immediate Post-test to Retention Test
Description: The official AHA Heartsave adult CPR AED Skill Sheet checklist for single-rescuer BLS was used to capture participants' skills for single-rescuer BLS and defibrillation with an AED. The AHA Heartsaver checklist has 11 action items, participant receives 1 point when an action on the checklist is performed. Therefore, the total score range from 0-11, with higher values represent a better outcome. Immediate post-test and retention test skill performance were evaluated by 2 independent raters. Skill retention was estimated by calculating the change in score from immediate post-test to retention test.
Time Frame: Baseline and 4 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Time Based | Mastery Based
Number analyzed (Participants) | 20 | 23
units on a scale
  Immediate post test total score | 8.0 [6.125 to 8.375] | 8.0 [7.0 to 9.0]
  Retention test total score | 8.5 [5.625 to 9.2] | 7.0 [6.0 to 8.0]

ADVERSE EVENTS:
Time Frame: Baseline to 4 months
Arm/Group | Time Based | Mastery Based
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/27
Other Adverse Events (participants affected / at risk) | 0/22 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No